CLINICAL TRIAL: NCT00382135
Title: An Evaluation of Semen Characteristics After 40 Weeks Daily Dosing With 20 mg Tadalafil
Brief Title: A Study of Semen Characteristics After 9 Months of Daily Tadalafil 20 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7011; H6D-MC-LVFE
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Erectile Dysfunction
Keywords: Impotence; erectile dysfunction; semen; sperm; Healthy male volunteers; men with mild erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo
- 2 (Active Comparator): 20 mg tadalafil tablet
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20mg tadalafil tablet taken by mouth once a day for 40 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: placebo — Placebo tablet taken by mouth once a day for 40 weeks
  Arms: 1

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, fixed dose, parallel design study to evaluate effects on semen characteristics after 40 weeks of daily dosing with 20 mg tadalafil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or men with mild erectile dysfunction
* At least 45 years of age
* With specified semen characteristics.

Exclusion Criteria:

* Certain chronic medical conditions including cardiac disease, congestive heart failure, kidney or liver disease, cancer and HIV
* A history of certain endocrine or hormonal abnormalities
* A history of significant testicular/genital abnormalities
* Any significant reproductive abnormality identified at the start of the study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-11; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in sperm production measured at baseline and after 9 months of treatment. | 40 weeks

SECONDARY OUTCOMES:
Changes in other semen characteristics and reproductive hormones. | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bothell, Washington, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com